CLINICAL TRIAL: NCT06729541
Title: Development and Application of Precision Treatment Strategies for Patients with Depression, Bipolar Disorder, and Schizophrenia: a Multicenter Randomized Controlled Trial
Brief Title: Development and Application of Precision Treatment Strategies for Common Mental Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Weihua Yue, Professor, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-23
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Depression - Major Depressive Disorder; Schizophrenia Disorders; Bipolar Disorder (BD)
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided (Experimental): In the Guided group, clinicians selected or maintained treatment based on patients' symptoms, incorporating pharmacogenomic testing. Patients underwent pharmacogenomic testing and received the results within 3 to 5 working days. Following this, drug dose adjustments or changes were made within the subsequent week (dose adjustments or changes were completed within 2 weeks of enrollment to ensure a stable dose). For schizophrenia (SCH), antipsychotic monotherapy was employed; for major depressive disorder (MDD), antidepressant monotherapy was initiated; and for bipolar disorder (BPD), mood stabilizer therapy was started with lithium or a single-agent valproic acid salt, along with regular monitoring of blood lithium levels. If symptoms remained uncontrolled after 2 to 4 weeks, consideration was given to adding a second mood stabilizer or psychiatric medication in combination with lithium or valproic acid salt.
  After 10 weeks of clinical observation, patients were assessed using standar
  Interventions: Other: Multigenetic Pharmacogenomics-Guided Treatment (MPGT)
- Unguided (No Intervention): In the Unguided group, clinicians selected or maintained treatment based on patients' symptoms, without the use of pharmacogenomic guidance. Patients underwent pharmacogenomic testing, and the results were provided at the end of the 12-week follow-up period. During the 12 weeks of clinical observation, patients were assessed using standardized scales at 4, 8, and 12 weeks. Clinical doctors adjusted the treatment plan based on the patients' clinical manifestations and assessment results at these intervals. The pharmacogenomic test report was delivered to patients at the conclusion of the 12-week follow-up period.

INTERVENTIONS:
Other: Multigenetic Pharmacogenomics-Guided Treatment (MPGT) — In the guidance group, drug types and dosages were adjusted based on the results of Pharmacogenetic TESTING.
  Arms: Guided

SUMMARY:
Schizophrenia (SCH), major depressive disorder (MDD), and bipolar disorder (BPD) are prevalent, disabling psychiatric conditions that not only cause significant suffering for affected individuals and their families but also impose a substantial socioeconomic burden and challenge societal well-being. Addressing the mental health challenges faced by patients, their families, and the healthcare system is a critical global public health priority. However, a comprehensive and systematic precision treatment approach for mental disorders remains largely absent in current clinical practice.

This study leveraged pharmacogenomic insights tailored specifically to the Chinese Han population to guide individualized medication selection. The approach incorporated quantitative assessment-based treatment protocols alongside therapeutic drug monitoring throughout the treatment process. The overarching goal was to establish a systematic precision treatment model that integrates "quantitative assessment-based treatment + pharmacogenomics + therapeutic drug monitoring." This model aims to optimize treatment outcomes, enhance safety, improve efficiency, and reduce costs, ultimately benefiting patients with psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia: (1) Age 18-65 years, no gender restriction, Han ethnicity; (2) Diagnosis confirmed using the MINI-International Neuropsychiatric Interview (MINI) tool, meeting the DSM-5 criteria for schizophrenia; (3) Baseline Positive and Negative Syndrome Scale (PANSS) score ≥ 60; (4) Education level of middle school or higher, no language barriers, able to cooperate with assessment and treatment, and informed consent obtained from the patient or guardian.
* Depressive Disorder: (1) Age 18-65 years, no gender restriction, Han ethnicity; (2) Diagnosis confirmed using the MINI tool, meeting the DSM-5 criteria for depressive disorder; (3) Baseline Hamilton Depression Rating Scale (HAMD-17) score ≥ 17; (4) Education level of middle school or higher, no language barriers, able to cooperate with assessment and treatment, and informed consent obtained from the patient or guardian.
* Bipolar Disorder: (1) Age 18-65 years, no gender restriction, Han ethnicity; (2) Diagnosis confirmed using the MINI tool, meeting the DSM-5 criteria for manic or hypomanic episodes in bipolar disorder; (3) Baseline Young Mania Rating Scale (YMRS) score ≥ 13; (4) Education level of middle school or higher, no language barriers, able to cooperate with assessment and treatment, and informed consent obtained from the patient or guardian.

Exclusion Criteria:

* Patients with a history of or currently meeting the DSM-5 criteria for the following diagnoses: organic mental disorders, schizoaffective disorder, intellectual disability, dementia, other cognitive disorders, alcohol or drug dependence, and Axis II disorders including personality disorders;
* Patients with severe suicidal tendencies (as assessed by the MINI Chinese version suicide module with a moderate risk or higher), or those at risk of harming others;
* Patients with severe or unstable physical illnesses;
* Narrow-angle glaucoma;
* A history of epilepsy or seizures;
* Known pregnancy and/or breastfeeding, or those planning to become pregnant;
* Participation in another clinical trial, or unwilling or unable to complete the full course of this trial;
* Participants deemed unsuitable by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) | Weeks 4, 8, and 12 of the treatment duration
  The outcome is assessed by the Positive and Negative Syndrome Scale (PANSS). The PANSS consists of 30 items, divided into three subscales: Positive Symptoms (7 items), Negative Symptoms (7 items), and General Psychopathology (16 items). Each item is rated on a 7-point scale from 1 (absent) to 7 (extreme), with higher scores indicating more severe symptoms. The total PANSS score ranges from 30 to 210, with higher scores reflecting greater symptom severity.
Change from baseline in Hamilton Depression Rating Scale (HAMD) | Weeks 4, 8, and 12 of the treatment duration
  The outcome is assessed by 17-item Hamilton Depression Rating Scale (HAMD-17) Scale. Total HAMD scores range from 0 to 24, with higher scores indicating more severe depressive symptoms.
Change from baseline in Young Mania Rating Scale (YMRS) | Weeks 4, 8, and 12 of the treatment duration
  The outcome is assessed by the Young Mania Rating Scale (YMRS). The YMRS consists of 11 items that assess the severity of manic symptoms, including mood, speech, motor activity, sexual interest, sleep, and other behaviors. Each item is rated on a scale from 0 to 4, with higher scores indicating greater severity of manic symptoms. The total YMRS score can range from 0 to 44, with higher scores reflecting more severe mania.

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | Weeks 4, 8, and 12 of the treatment duration
  The outcome is assessed by the Clinical Global Impression (CGI) scale. The CGI consists of two main components: the CGI-Severity (CGI-S) and the CGI-Improvement (CGI-I).
  CGI-Severity (CGI-S): This component rates the severity of the patient's illness on a 7-point scale, ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  CGI-Improvement (CGI-I): This component evaluates the patient's improvement over time, also on a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse).
  The CGI scale provides an overall clinical assessment of the patient's condition, considering both the severity of illness and the degree of improvement.
Morisky Medication Adherence Scale (MMAS) | Weeks 4, 8, and 12 of the treatment duration, as well as Months 6 and 12.
  The outcome is assessed by the Morisky Medication Adherence Scale (MMAS). The MMAS is a self-reported scale used to assess a patient's adherence to prescribed medication regimens. It consists of 8 items that evaluate factors such as forgetfulness, understanding of medication instructions, and attitude toward treatment. The items are answered with "yes" or "no" responses, with higher scores indicating better medication adherence.
  The MMAS is categorized as follows:
  High adherence: score of 8 Medium adherence: score of 6-7 Low adherence: score of 0-5
Plasma Drug Concentration | Weeks 4, 8, and 12 of the treatment duration
  The outcome is assessed by Plasma Drug Concentration. Blood drug levels of antidepressants, antipsychotics, and mood stabilizers are measured to determine whether the concentrations fall within the therapeutic range for each respective medication. Therapeutic drug monitoring ensures that plasma drug levels are within the safe and effective range, avoiding both sub-therapeutic and potentially toxic concentrations. The concentration of each drug is compared to the recommended therapeutic window to assess if the patient is receiving an optimal dose.
Personal and Social Performance Scale (PSP) | Weeks 4, 8, and 12 of the treatment duration, as well as Months 6 and 12.
  The outcome is assessed by the Personal and Social Performance Scale (PSP). The PSP is a clinician-rated scale designed to assess an individual's level of functioning in four key areas:
  Socially useful activities (e.g., work, education, social relationships) Personal and social relationships (e.g., relationships with family, friends, and the community) Self-care (e.g., personal hygiene, ability to live independently) Disturbing and aggressive behavior (e.g., level of agitation or violence)
  The PSP provides a global score ranging from 1 to 100, where lower scores indicate more severe dysfunction and higher scores indicate better social and personal performance. The total PSP score is classified as follows:
  Score 91-100: Normal functioning Score 61-90: Mild functional impairment Score 31-60: Moderate functional impairment Score 1-30: Severe functional impairment
Safety | Weeks 4, 8, and 12 of the treatment duration
  Laboratory tests (including complete blood count, liver and kidney function, prolactin levels, and electrocardiogram) were conducted at baseline and at Weeks 4, 8, and 12 of the treatment duration. Safety was assessed using adverse event scales (e.g., TESS and SAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hostipal, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No